CLINICAL TRIAL: NCT03170830
Title: Study on CircRNA-Uck2 as a New Diagnostic Marker of Acute Myocardial Infarction
Brief Title: Diagnostic Value of CircRNA-Uck2 for Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Haidian Hospital (Other)
Collaborators: Beijing Fangshan District Liangxiang Hospital (Other)
Responsible Party: Principal Investigator, Hong-Jin Wu, Clinical Professor, Beijing Haidian Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KYZ2017001
Record Dates: First submitted 2017-05-19; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cardiac Disease; Diagnoses Disease; Acute Myocardial Infarction
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sample inspector
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control group (Experimental): Age:45-75 years.Pepole who have normal ECG without the history of cardiovascular disease can be included in the healthy control group.
  Interventions: Diagnostic Test: the diagnosis value of cUck2 in acute myocardial infarction.
- unstable angina disease control group (Experimental): Age:>18 years.Unstable angina patients meet the diagnostic criteria.
  Interventions: Diagnostic Test: the diagnosis value of cUck2 in acute myocardial infarction.
- acute myocardial infarction group (Experimental): Age:>18 years.Acute myocardial infarction patients meet the diagnostic criteria.
  Interventions: Diagnostic Test: the diagnosis value of cUck2 in acute myocardial infarction.

INTERVENTIONS:
Diagnostic Test: the diagnosis value of cUck2 in acute myocardial infarction. — Collect blood at different time points and compare cUck2 in three groups.

SUMMARY:
This is an observational diagnostic study that aims to evaluate the diagnostic value of circRNA-Uck2 in Acute Myocardial Infarction (AMI) in adults as compared to healthy and unstable angina controls. Rapid and adequate diagnosis of AMI is of great importance to enable a rapid start of treatment, save large tracts of dying myocardium, reduce the infarct size,and thereby decrease the risk of subsequent heart failure.

DETAILED DESCRIPTION:
RATIONAL acute myocardial infarction (AMI) is the leading cause of sudden death and heart failure worldwide. And about 10% of all emergency department consultations are with symptoms suggestive of AMI, however, only 10% to 20% of them are diagnosed as experiencing an AMI. Rapid and accurate identification of AMI is of paramount clinical importance for subsequent timely and effectively treatment and management.

Recently, the investigators identified microarray analysis and real-time polymerase chain reaction (PCR) from AMI animal models and small samples of AMI patients, a molecular signature of AMI involving 5 circRNAs (circRNA_006877, circRNA_015350, circRNA_002969, circRNA_013240, circRNA_004682) was found significantly change in AMI patients and likely serves as candidate serum biomarkers of AMI. Among the 5 circRNAs, circRNA_006877 name of circRNA-Uck2 (cUck2) has more close association with AMI.

TYPE OF STUDY : multicenter diagnostic evaluation Study MAIN PURPOSE OF THE STUDY : To evaluate the diagnostic value of circRNAs in AMI in adults as compared to healthy and unstable angina controls

SECONDARY OBJECTIVES :

assess the ability of cUck2 to discriminate a AMI disease from unstable angina patients in adults.

explore the relationship between cUck2 and heart function after myocardial infarction PRODUCTS OF THE STUDY diagnostic kit of AMI in quantitative polymerase chain reaction (qPCR) NUMBER OF PATIENTS : 3 groups with 169 patients will be included Group 1: 66 AMI adult patients Group 2: 56 unstable angina adults Group 3: 56 Witnesses healthy adults INCLUSION LENGTH 36 months DURATION OF THE STUDY 42 months

ELIGIBILITY:
Inclusion Criteria:

* Health Control Group:Pepole who have normal ECG, deny the history of cardiovascular disease can be included in the healthy control group.
* Acute Myocardial Infarction Group:Clinical diagnosis of acute myocardial infarction
* Unstable Angina Group:Clinical diagnosis of unstable angina.
* Sign informed consent.

Exclusion Criteria:

* Myocarditis, hypertrophic cardiomyopathy, ablation.
* Malignant hypertension, severe arrhythmia.
* Chronic muscle disorders, rhabdomyolysis.
* Severe liver and kidney dysfunction.
* Malignant tumors, acute cerebrovascular disease.
* Severe neurosis, psychosis.
* Patients who had any of the above were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The change of cUck2 levels in AMI | It is totally 7 time points to detect cUck2, including the moment of admission, and the 1st day、the 2nd day、the 3th day、the 7th day、the 14th day、the 6th month after admission in AMI patients.
  The investigators has found cUck2 has more close association with AMI.Detect cUck2 levels in different time points and it will give more information about its diagnostic value in AMI.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Jin Wu, Study Director — Beijing Haidian Hospital,Haidian Section of Peking University Third Hospital
Locations (1):
- Beijing Haidian Hospital, Haidian Section of Peking University Third Hospital, Beijing, China/Beijing, China

REFERENCES:
- [Background] Danese E, Montagnana M. An historical approach to the diagnostic biomarkers of acute coronary syndrome. Ann Transl Med. 2016 May;4(10):194. doi: 10.21037/atm.2016.05.19. PMID 27294090
- [Background] Sanger HL, Klotz G, Riesner D, Gross HJ, Kleinschmidt AK. Viroids are single-stranded covalently closed circular RNA molecules existing as highly base-paired rod-like structures. Proc Natl Acad Sci U S A. 1976 Nov;73(11):3852-6. doi: 10.1073/pnas.73.11.3852. PMID 1069269
- [Background] Jeck WR, Sorrentino JA, Wang K, Slevin MK, Burd CE, Liu J, Marzluff WF, Sharpless NE. Circular RNAs are abundant, conserved, and associated with ALU repeats. RNA. 2013 Feb;19(2):141-57. doi: 10.1261/rna.035667.112. Epub 2012 Dec 18. PMID 23249747
- [Background] Suzuki H, Zuo Y, Wang J, Zhang MQ, Malhotra A, Mayeda A. Characterization of RNase R-digested cellular RNA source that consists of lariat and circular RNAs from pre-mRNA splicing. Nucleic Acids Res. 2006 May 8;34(8):e63. doi: 10.1093/nar/gkl151. PMID 16682442
- [Background] Holdt LM, Stahringer A, Sass K, Pichler G, Kulak NA, Wilfert W, Kohlmaier A, Herbst A, Northoff BH, Nicolaou A, Gabel G, Beutner F, Scholz M, Thiery J, Musunuru K, Krohn K, Mann M, Teupser D. Circular non-coding RNA ANRIL modulates ribosomal RNA maturation and atherosclerosis in humans. Nat Commun. 2016 Aug 19;7:12429. doi: 10.1038/ncomms12429. PMID 27539542
- [Background] Wang K, Long B, Liu F, Wang JX, Liu CY, Zhao B, Zhou LY, Sun T, Wang M, Yu T, Gong Y, Liu J, Dong YH, Li N, Li PF. A circular RNA protects the heart from pathological hypertrophy and heart failure by targeting miR-223. Eur Heart J. 2016 Sep 1;37(33):2602-11. doi: 10.1093/eurheartj/ehv713. Epub 2016 Jan 21. PMID 26802132
- [Background] Meder B, Keller A, Vogel B, Haas J, Sedaghat-Hamedani F, Kayvanpour E, Just S, Borries A, Rudloff J, Leidinger P, Meese E, Katus HA, Rottbauer W. MicroRNA signatures in total peripheral blood as novel biomarkers for acute myocardial infarction. Basic Res Cardiol. 2011 Jan;106(1):13-23. doi: 10.1007/s00395-010-0123-2. Epub 2010 Oct 1. PMID 20886220